CLINICAL TRIAL: NCT07160166
Title: Determination of the Oral Irritation Potential of Two Alcohol-Free Rinses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kenvue Brands LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS2025OC100242
Record Dates: First submitted 2025-07-22; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Oral Health

STUDY DESIGN:
Intervention Model Description: This is a single center, examiner-blind, randomized, parallel-group, controlled clinical trial.
Who Masked: Investigator
Masking Description: Examiner-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Prototype 1 Regimen (Experimental): All subjects will receive a marketed fluoride-containing dentifrice (Colgate® Cavity Protection) and a soft flat trimmed bristled toothbrush and their assigned mouthwash at their Screening/Baseline visit to use throughout the study. Subjects will use their assigned study products and complete their oral care regimen for the first time at the site under supervision. At home, subjects will brush twice daily for at least 1 timed minute with the toothpaste and toothbrush provided. After brushing for at least 1 timed minute, subjects will rinse with their assigned mouthwash according to the product label. Subjects will be required to record their twice daily product usage on a subject diary starting with their first product use at the site.
  Interventions: Other: Prototype 1
- Experimental: Prototype 2 Regimen (Experimental): All subjects will receive a marketed fluoride-containing dentifrice (Colgate® Cavity Protection) and a soft flat trimmed bristled toothbrush and their assigned mouthwash at their Screening/Baseline visit to use throughout the study. Subjects will use their assigned study products and complete their oral care regimen for the first time at the site under supervision. At home, subjects will brush twice daily for at least 1 timed minute with the toothpaste and toothbrush provided. After brushing for at least 1 timed minute, subjects will rinse with their assigned mouthwash according to the product label. Subjects will be required to record their twice daily product usage on a subject diary starting with their first product use at the site.
  Interventions: Other: Prototype 2
- Active Comparator: Marketed Comparator Regimen (Active Comparator): All subjects will receive a marketed fluoride-containing dentifrice (Colgate® Cavity Protection) and a soft flat trimmed bristled toothbrush and their assigned mouthwash at their Screening/Baseline visit to use throughout the study. Subjects will use their assigned study products and complete their oral care regimen for the first time at the site under supervision. At home, subjects will brush twice daily for at least 1 timed minute with the toothpaste and toothbrush provided. After brushing for at least 1 timed minute, subjects will rinse with their assigned mouthwash according to the product label. Subjects will be required to record their twice daily product usage on a subject diary starting with their first product use at the site.
  Interventions: Other: Marketed Comparator

INTERVENTIONS:
Other: Prototype 1 — Subjects will brush and rinse with their assigned mouthwash twice daily.
  Arms: Experimental: Prototype 1 Regimen
Other: Prototype 2 — Subjects will brush and rinse with their assigned mouthwash twice daily.
  Arms: Experimental: Prototype 2 Regimen
Other: Marketed Comparator — Subjects will brush and rinse with their assigned mouthwash twice daily.
  Arms: Active Comparator: Marketed Comparator Regimen

SUMMARY:
The objective of this study is to evaluate the oral soft and hard tissue tolerance after 14 days of a twice daily regimen of brushing and rinsing with essential oil containing alcohol free mouthwashes versus a control.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 18 years of age and older, at the time of screening/baseline (approximately 15% Black and 5% Asian race; approximately 10% Hispanic ethnicity).
2. Generally, in good general and oral health (i.e. brush teeth daily and exhibit no signs of gross oral neglect) without any known allergy to commercial dental products or cosmetics.
3. Able to comprehend and follow the requirements and restrictions of the clinical trial (including willingness to use the assigned study products per instructions, availability on scheduled visit dates and likeliness of completing the clinical trial) based upon research site personnel's assessment.
4. Individual has signed the Consent for Photograph Release and ICD (and/or Assent Document, as applicable)including Health Insurance Portability and Accountability Act (HIPAA) disclosure.
5. Able to read and understand the local language (subject is capable of reading the documents).
6. Generally, in good health based on medical history reported by the subject.
7. In good oral health with adequate oral hygiene (i.e. brush teeth daily and exhibit no signs of gross oral neglect).
8. Negative pregnancy urine tests (females of child-bearing potential only):

   * For females: Postmenopausal state (i.e. at least 1 year without menses without an alternative medical condition prior to the first study IP administration) or premenopausal/perimenopausal state with an effective means of contraception.
   * For males: No pregnant or lactating spouse or partner at screening and willingness to utilize an acceptable form of birth control with spouse or any potential partner during the study and for 30 days thereafter.
9. Females of childbearing potential must be using a medically acceptable method of birth control for at least one month prior to Visit 1 and agree to continue using this method during their participation in the clinical trial. Medically acceptable forms of birth control that may be used by the subject and/or his/her partner include:

   * Double barrier method (condoms, diaphragm or cervical cap with spermicide),
   * Hormonal prescription contraceptives (i.e., oral, injectable, implanted, patch or vaginal ring hormone therapy)
   * Intrauterine device (IUD)
   * Surgical sterilization (e.g., vasectomy that has been confirmed effective by sperm count check, tubal ligation, hysterectomy and/or bilateral oophorectomy)
   * Abstinence
10. A minimum of 16 uncrowned teeth.
11. Absence of significant oral soft tissue pathology, periodontitis and active dental caries, based on a visual examination and at the discretion of the Investigator.
12. Absence of partial dentures, dentures, orthodontic bands, fixed retainers, removable orthodontic appliances.

Exclusion Criteria:

1. Diagnosed with Xerostomia.
2. Suspected alcohol or substance abuse at the discretion of the Investigator (e.g., amphetamines, benzodiazepines, cocaine, marijuana, opiates).
3. Known sensitivity, allergy or contraindications to any investigational product ingredient, oral care products and auxiliary supplies provided for the study.
4. Self-reported smokeless tobacco user including snuff, chewing tobacco, vaping and e-cigarette usage.
5. Females who are self-reported to be pregnant, planning to become pregnant or breastfeeding during the study.
6. Participation in any clinical study investigation within 30 days of Screening visit (Visit 1).
7. Planned surgery during the trial period, 6 months prior to clinic visit 1 or 30 days after the end of study period.
8. Has a compromised immune system, in the judgement of the medically qualified investigator.
9. Has any acute or chronic, medical or psychiatric conditions) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgement of the medically qualified investigator, would make the subject inappropriate for entry in this study;
10. Significant, unstable or uncontrolled medical condition which may interfere with subject's participation in the study, at the discretion of the Investigator.
11. Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication;
12. Is taking a medication that would mask an Adverse Event (AE) or confound the study results, including:

    * Immunosuppressive or steroidal drugs within 2 months before Visit 1.*
    * Non-steroidal anti-inflammatory drugs within 5 days before Visit 1.
    * Antihistamines within 2 weeks before Visit 1.
13. Subjects who are related to those persons involved directly or indirectly with the conduct of this study (i.e., principal Investigator, sub-investigators, study coordinators, other site personnel, employees of Kenvue Brands LLC/Johnson & Johnson (J&J) subsidiaries, contractors of Kenvue/J&J, and the families of each).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2025-07-11 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Change in baseline in oral tolerance based on oral hard and soft tissue exams | Up to Day 14
  Change in baseline in oral tolerance based on oral hard and soft tissue exams will be reported. Oral examinations will be conducted to monitor oral hard and soft tissues tolerance to the treatments. Buccal and sublingual mucosae, lips/labial mucosa, mucobuccal gold, gingiva, tongue, hard and soft palate, uvula, oropharynx, teeth and dental restorations will be examined and findings will be recorded in the electronic data capture (EDC) system.
Number of Participants with Adverse Events (AEs) | Up to Day 14
  An AE is any untoward medical occurrence in a clinical study participant temporarily associated with the clinical investigation, whether or not the event has a causal relationship to the participant's participation in the trial.

SECONDARY OUTCOMES:
Mouthwash Habits Baseline Questionnaire | Visit 1 (Day 0)
  For the Mouthwash Habits Baseline Questionnaire, the number and percentage of subjects for each response of each question will be presented by investigational product group. For these aggregated response categories, percentages of subjects will be compared between investigational product groups using a chi-square test, or Fisher's exact test if the expected cell size is sufficiently small.
  For ordinal response questions (9-point Liking scales and 5-point scales), the mean and standard deviation for each ordinal response variable will also be displayed.
  Each statistical test will be carried out at the 0.10 level of significance, two-sided. Note that testing at the 0.10 level of significance is reasonable for consumer perception testing, as decisions based on these types of data are typically based on this significance level.
Product Perception Claims Questionnaire | Visit 3 (Day 14 ± 1 day)
  For the Product Perception Claims Questionnaire, the number and percentage of subjects for each response of each question will be presented by investigational product group.
  For these aggregated response categories, percentages of subjects will be compared between investigational product groups using a chi-square test, or Fisher's exact test if the expected cell size is sufficiently small.
  For ordinal response questions (9-point Liking scales and 5-point scales), the mean and standard deviation for each ordinal response variable will also be displayed.
  Each statistical test will be carried out at the 0.10 level of significance, two-sided. Note that testing at the 0.10 level of significance is reasonable for consumer perception testing, as decisions based on these types of data are typically based on this significance level.
Comparison of the salivary microbial counts | Visit 1 (Day 0); Visit 3 (Day 14 ± 1 day)

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No